CLINICAL TRIAL: NCT06698627
Title: IMPRIVE Pilot Study: Comparison of Two Over the Counter Intravaginal Devices for the Treatment of Stress Urinary Incontinence
Brief Title: Comparison of Two Over the Counter Intravaginal Devices for the Treatment of Stress Urinary Incontinence
Acronym: IMPRIVE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Elisabeth Sebesta, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 23113
Record Dates: First submitted 2024-11-18; First posted 2024-11-21 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Stress Urinary Incontinence in Women
Keywords: stress urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: Prior to randomization participants will be sent the Poise Impressa sizing kit via mail. They will then be asked what size of device works best for them based on the sizing kit. After this information is obtained they will then be sent both Revive and correct size of Poise Impressa. They will be randomized at this time regarding which device they will start with. If participants are menstruating, they will be asked to start this study after their last day of bleeding as this study will last approximately 20 days. They will then begin using the device they were randomized to use first for 7 days. There will be a three day wash out period and them they will use the remaining device for 7 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Poise Impressa (Active Comparator): Participants will be asked to use Poise Impressa for 7 days based on package insert
  Interventions: Device: Daily Disposable Continence Device
- Revive (Active Comparator): Participants will be asked to use Revive continence device based on package insert.
  Interventions: Device: Monthly Disposable Continence Device

INTERVENTIONS:
Device: Daily Disposable Continence Device — The Poise® Impressa® is an over-the-counter intravaginal device for women over the age of 21 years with SUI. It is a disposable, one-time use tampon-like device that comprises a core, cover, and applicator. The device is inserted and removed like a vaginal tampon and comes in three sizes.
  Arms: Poise Impressa
Device: Monthly Disposable Continence Device — The Revive® is another over the counter vaginal insert for the treatment of SUI. This is a self-deployable, double-loop pessary device.
  Arms: Revive

SUMMARY:
The goal of this pilot study is to compare two commercially available over the counter devices for treatment of stress urinary incontinence in a web based format.

The main questions it aims to answer

1. What device do women with SUI prefer after using both devices
2. What patient factors help drive this preference if any
3. Is a web-based crossover intervention study feasible

Participants will:

Use two over the counter devices over a course of 20 days. They will have both devices sent via mail.

They will answer questions prior to the start of using any device and then after using each device They will be asked to complete daily bladder diaries

DETAILED DESCRIPTION:
Pelvic floor disorders (PFD) are common in the United States with an estimated 25% of women experiencing one of more pelvic floor disorder. PFDs include pelvic organ prolapse (POP), urinary incontinence (UI), and fecal incontinence (FI). These disorders have been associated with significant distress. Treatment options include both surgical and non-surgical management. Non-surgical options for treatment of stress urinary incontinence (SUI) include pelvic floor physical therapy, pessary, and over-the counter vaginal insertion devices. The Poise® Impressa® is an over-the-counter intravaginal device for women over the age of 21 years with SUI. It is a disposable, one-time use tampon-like device that comprises a core, cover, and applicator. The device is inserted and removed like a vaginal tampon and comes in three sizes. In an open-label controlled study, 60 women with severe urodynamic stress incontinence tested the device for 28 days. 85% of participants achieved a greater than 70% reduction in pad weight gain, and mean pad weight gain decreased from 17g per 8 hours to 2 g per 8 hours. A high degree of satisfaction was reported, and 70% of participants reported 90% improvement (Ziv et al). The Revive® is another over the counter vaginal insert for the treatment of SUI. This is a self-deployable, double-loop pessary device. (Ziev et al) conducted a multicenter, interventional, single-arm study and found 71% of the study population experienced a >50% reduction in leakage volume, leakage episodes, or both. Participants quality-of-life scores improved from baseline to post treatment phase by 4.35 points on average (p<0.0001).

Although over the counter vaginal inserts are a treatment option for SUI, it is not known if patients that are evaluated by medical practitioners are presented with this as a treatment as part of conservative management. The most recent Cochrane review on mechanical devices for the management of UI (Lipp et al., 2014) summarized the results of eight randomized trials reflecting the use of standard available intravaginal pessaries, tampons, and other intravaginal and intraurethral devices. As most trials were small, outcome measures were diverse, and few trials included control/no-treatment groups, the data regarding the use of mechanical devices for treatment of UI are still unclear. Additionally, some of these products are recommended in office by providers without current robust data regarding patient reported outcomes. The available data is limited to safety/efficacy data supported by the manufacturers of these devices. Ideally, this work could inform counseling and recommendations for providers that evaluate patients for stress urinary incontinence. For example, a subset of women that present for evaluation in clinic desire to proceed with surgical correction for SUI with urethral bulking or sling. In the interim prior to their scheduled surgery often only hygiene products can be offered that do not address the cause of leaking. Additionally, the market for these products is large and it is unclear how different women are experiencing these products. It is important to collect demographic information on who these products may be working the best for. This pilot project can help to collect some of these demographic information. Furthermore, there are a significant amount of women across the United States that do not have access to subspeciality urogynecologist or female urologists and use these devices without ever interacting with the healthcare system or getting a specific recommendation. For these women it is important that data exists from which they determine which of the commercially available devices may work best for them and may be more effective/affordable. Ultimately, this study will be helpful in determining the feasibility of the online format for this type of study. Also, once completed the information collected in this study could help to generate multiple hypotheses for larger confirmatory studies. Thus, further investigation into these treatment options is warranted. To date, no comparative trials have been performed to compare the Revive and the Impressa over the counter vaginal inserts in women seeking non-operative therapy for SUI. The investigators aim to perform a cross-over comparative effectiveness trial to evaluate SUI treatment success using two OTC vaginal inserts currently commercially available.

Prior to randomization participants will be sent the Poise Impressa sizing kit. Participants will then be asked what size of device works best for them based on the sizing kit. After this information is obtained that will then be sent both Revive and correct size of Poise Impressa. Participants will be randomized at this time. If participants are menstruating, participants will be asked to start this study after their last day of bleeding as this study will last approximately 20 days.

Example of participant timeline assuming randomized to Revive device first

Day 1-3

* Participant will perform ICIQ-SF, UDI-6, Incontinence Impact questionnaire (IIQ-7), Sandvik Severity Index
* Daily record of incontinence episode diary including number of pads used for incontinence

Week 1 (days 4-10)

* Revive® device
* UDI-6,IIQ-7, Sandvik severity index, ICIQ-SF)
* Device favorability score
* Patient global Impression of Improvement scale
* Daily record of incontinence episodes diary
* Satisfaction with device/comfort/success

Days (11-13) Three day wash out period with no incontinence device used

Week 2 (Days 14-20)

* Impressa® Device
* UDI-6, IIQ-7, Sandvik severity index, ICIQ-SF)
* Device favorability score
* Patient global Impression of Improvement scale
* Daily incontinence episodes diary
* Satisfaction with device/comfort/success

Statistical Analysis:

With planned enrollment of 80 patients and assuming a 20% dropout rate which is conservative compared to existing literature (McKay, H. Garth, et al), the investigators anticipate to have N=64 participants complete the study and provide rating for both device.

Sample size and estimates precision analysis The primary study end point will be the participants' preference on each device measured with a 5-level likert scale (Very favorable, favorable, neutral, unfavorable, or very unfavorable). The investigators conducted a simulation study with 64 participants (32 per sequence arm). In this simulation, the investigators assumed that participants were 20% more likely to choose Favorable/Very favorable for Impressa than for Revive. The results from a series of scenarios suggest that 60.9% of time, participants will prefer Impressa over Revive (by comparing the 5-lever likert scale), with a 95% confidence interval of 50% to 71.1% (assume 70% vs. 50% choose Favorable/Very favorable for the two devices respectively).

Statistical Analysis Plan All participants characteristics will be summarized using median with interquartile range (for continuous variables) and frequency with percentage (categorical variables). In the primary analysis, to allow the tie of rating for the two devices, the investigators will use the Prescott test to evaluate the difference of device preference measured by the 5-level likert scale (the primary endpoint). In a secondary analysis, the investigators will analyze the participants' rating for both devices as an ordinal outcome. The investigators will use ordinal regression models while taking into consideration the potential unbalanced participants characteristics. The investigators believe that the washout period used in this study is sufficient and carryover effect is unlikely.

ELIGIBILITY:
Inclusion Criteria:

Women with a history of stress urinary incontinence that have not undergone treatment that desire conservative management.

Inclusion criteria:

* 21 years or older
* Patients will be screened for inclusion criteria using the MESA. This questionnaire helps to identify patients with mixed urinary incontinence (MUI) and help distinguish between stress predominant mixed urinary incontinence and urge predominant mixed urinary incontinence. The UUI score should be zero. We will not allow patients that have MUI to be included in the study based on the MESA.
* Report an average loss of urine greater than three episodes per week.
* Ability to receive mail through USPS

Exclusion Criteria:

* Patient should not be on vacation at time of study and should be performing daily activities.
* Inability to follow packaged instructions for insertion devices chosen to be included within this study
* Pregnancy or plan to become pregnant in the next three months
* Significant vaginal atrophy due to genitourinary syndrome of menopause
* Current use of over-the-counter vaginal insertion device for treatment of stress urinary incontinence
* Post-menopausal bleeding
* Participants that report visible prolapse and/or bother symptoms of prolapse
* Bladder modifying medications
* Unable to use incontinence device per package instructions
* Given birth in the past three months
* Had vaginal surgery in the last three months
* IUD placement in the past 6 months
* Vaginal infection or UTI that is active
* Undergoing pelvic floor physical therapy
* Had vaginal surgery within the last three months

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Device Preference | Day 10, Day 20
  Women will be asked to rate each device on a 5 point Likert scale of 1-5.
  The options for responses will include very favorable, favorable, neutral, unfavorable, very unfavorable. The response for each device will then be compared.

SECONDARY OUTCOMES:
Patient's global improvement in urinary incontinence | Day 10 and Day 20
  The PGI-I is a validated questionnaire assessing a patient's global improvement in urinary incontinence following a specific intervention on a 7-item Likert scale including "very much better," "much better," "a little better," "no change," "a little worse," "much worse" and "very much worse."
  Responses of much better or very much better will be determined as treatment success.
  The Patient Global Impression of Severity and of Improvement question responses were correlated significantly with incontinence episode frequency, stress pad test, and Incontinence Quality of Life Questionnaire measures, which established the construct validity of these two global assessment questions for baseline severity and treatment response, respectively.
Comparison of reduction in number incontinence episodes | Daily for 20 days
  Daily Bladder Diary. Participants will be asked the number of times they leaked in the day.
Comparison of symptom bother ICIQ-SF | Day 1, Day 10, Day 20
  The ICIQ-UI Short Form is a questionnaire for evaluating the frequency, severity and impact on quality of life (QoL) of urinary incontinence in men and women in research and clinical practice across the world. This short and simple questionnaire is also of use to general practitioners and clinicians in both primary and secondary care institutions to screen for incontinence, to obtain a brief yet comprehensive summary of the level, impact and perceived cause of symptoms of incontinence and to facilitate patient-clinician discussions.
  Scoring is from 0-21. The higher the score the worse impact the patient symptoms has on quality of life.
Device Satisfaction | Day 10 and Day 20
  Satisfaction with device will be assessed using likert scale questionnaires assessing device satisfaction with the question and answers below.
  "How satisfied were you with the device?"
  Participants can select: ("somewhat satisfied" and "not at all satisfied" and very satisfied)
Device Comfort | Day 10 and Day 20
  Comfort of device will be assessed using likert scale questionnaires assessing device comfort
  In general, how comfortable was the device?"
  ("somewhat comfortable" and "not at all comfortable", completely comfortable)
Ease of use | Day 10 and Day 20
  Ease of use with device will be assessed using likert scale questionnaires assessing ease of use with the below question and answer.
  How easy/difficult was the device to use?"
  ("very easy", "easy", "neutral or unsure," , "difficult" , "very difficult")
Comparison of symptom bother UDI-6 | Day 1, Day 10, Day 20
  Urinary Distress Inventory (UDI-6): 6 questions measuring urinary incontinence symptom bother. Scale: 0-600.
  Having higher scores indicate higher level of bother.
Quality of Life Measure IIQ-7 | Day 1, Day 10, Day 20
  Incontinence Impact Questionnaire (IIQ-7): 7 questions measuring functional impact of urinary incontinence. Scale: 0-100.
  Having higher scores indicate higher level of bother.
Sandvik Severity Index | Day 1, Day 10, Day 20
  The Sandvik test was developed by Sandvik et al to be used as a simple way to calculate severity of urinary incontinence in women. According to the Sandvik index, women with a score of 1-2 are classified as mild incontinece severity, a score of 3-4 is classified as moderate, and a score of 6 or more is classified as severe.

OTHER OUTCOMES:
Continued patient product used after completion of study period | 3 months after intervention completion
  Participants will be asked if they can be contacted at the conclusion of the study. IF the participant agrees they will be contacted approximately 3 months after study completion to determine if patients continued to use one or both of the devices. Patients will also be asked if they decided to purchase any of the devices or went on to proceed with another treatment for SUI.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McKay HG, King D, Eakin EG, Seeley JR, Glasgow RE. The diabetes network internet-based physical activity intervention: a randomized pilot study. Diabetes Care. 2001 Aug;24(8):1328-34. doi: 10.2337/diacare.24.8.1328. PMID 11473065
- [Result] Nekkanti S, Wu JM, Hundley AF, Hudson C, Pandya LK, Dieter AA. A randomized trial comparing continence pessary to continence device (Poise Impressa(R)) for stress incontinence. Int Urogynecol J. 2022 Apr;33(4):861-868. doi: 10.1007/s00192-021-04967-9. Epub 2021 Sep 9. PMID 34505171
- [Result] Yalcin I, Bump RC. Validation of two global impression questionnaires for incontinence. Am J Obstet Gynecol. 2003 Jul;189(1):98-101. doi: 10.1067/mob.2003.379. PMID 12861145
- [Result] Duenas-Garcia OF, Shapiro RE, Gaccione P. Safety and Efficacy of a Disposable Vaginal Device for Stress Urinary Incontinence. Female Pelvic Med Reconstr Surg. 2021 Jun 1;27(6):360-364. doi: 10.1097/SPV.0000000000000861. PMID 32453209
- [Result] Ziv E, Stanton SL, Abarbanel J. Significant improvement in the quality of life in women treated with a novel disposable intravaginal device for stress urinary incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Jun;20(6):651-8. doi: 10.1007/s00192-009-0824-y. Epub 2009 Mar 11. PMID 19434384
- [Result] Ziv E, Stanton SL, Abarbanel J. Efficacy and safety of a novel disposable intravaginal device for treating stress urinary incontinence. Am J Obstet Gynecol. 2008 May;198(5):594.e1-7. doi: 10.1016/j.ajog.2008.01.061. Epub 2008 Apr 2. PMID 18377862
- [Result] Lipp A, Shaw C, Glavind K. Mechanical devices for urinary incontinence in women. Cochrane Database Syst Rev. 2014 Dec 17;2014(12):CD001756. doi: 10.1002/14651858.CD001756.pub6. PMID 25517397